CLINICAL TRIAL: NCT07102264
Title: Safety & Feasibility of Ultrasound-assisted Non-invasive Measurement of Compressibility of the Thyroid Gland in Patients Scheduled for Surgical Removal (CPMX-Thyr)
Brief Title: Safety & Feasibility of Ultrasound-assisted Non-invasive Measurement of Compressibility of the Thyroid Gland in Patients Scheduled for Surgical Removal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CPMX-Thyr
Record Dates: First submitted 2025-06-18; First posted 2025-08-03 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Nodule (Diagnosis)
MeSH Terms: conditions — Thyroid Nodule; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPMX1 measurement (Experimental): Measurement using investigational device CPMX 1 in addition to standard of care ultrasound.
  Interventions: Device: CPMX1

INTERVENTIONS:
Device: CPMX1 — Compressibility of thyroid nodules using CPMX1 during pre surgery planning visit

SUMMARY:
The thyroid gland plays an important role in hormone regulation however, it is often prone to nodules. This is common with nodules being found in up to 68% of people in a neck ultrasound, with likelihood increasing with age. However, only about 1 in 20 nodules turns out to be cancerous.

Diagnosis of thyroid nodules starts with ultrasonic assessment, where specific features have been identified to estimate the risk of malignancy. If further examination is recommended, Fine Needle Aspiration (FNA) is performed. A needle is inserted into the nodule and the obtained subset of cells are then classified into 6 categories (Bethesda score) after examination under the microscope. While some Bethesda scores provide very accurate malignancy predictions, others like category 4, are unspecific, with risk of malignancy ranging from 25 to 40%. For these patients, about 75% are operated on even though they are not prospectively diagnosed.

Soft tissue has certain physical properties, including its compressibility, which could be quantified by measuring the pressure required to deform it. It has been found that cancerous tissue is often harder than the surrounding healthy tissue. Compremium, a Swiss company which has its headquarters in Muri bei Bern, has developed a device that can be used to measure the compressibility of tissue, similarly to palpation but providing a quantitative assessment. The present study aims to investigate the feasibility and preliminary efficacy of this new technology to predict if thyroid nodules of patients scheduled for surgical removal based on FNA analysis are malignant or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with a thyroid node
* Patients with a Bethesda IV cytopathological diagnosis of this node
* Informed consent documented by signature

Exclusion Criteria:

* Non-intact skin at the measurement site
* BMI>35kg/m2
* Patients unable to provide informed consent
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Device safety | up to 6 months
  - The practitioner will be asked to identify any new risks arising during the measurements using the investigational device and report these in the CRF.
Device safety | Up to 6 months
  Safety of the device shall be evaluated by systematically reporting device deficiencies (DDs), adverse device events (ADEs) and Serious adverse device events (SADEs) and by monitoring the frequency and incidence of these events.
Device safety | Up to 6 months
  The participant will be asked to rate the perceived pain scale after the examination with the investigational device using a patient questionaire (Numeric Rating Scale).

SECONDARY OUTCOMES:
Preliminary efficacy of CPMX1 compressability values to predict thyroid nodule malignancy. | 60 minutes
  Preliminary efficacy of compressibility values measured with the thyroid investigational system to predict a thyroid nodule's malignancy will be assessed by:
  1. Computing discriminative ability and breaking down predictions into true and false positives and negatives
  2. Quantification of the prospective number of surgeries if compressibility were used for clinical decision making.
  The thyroid's malignancy prediction will be determined by using the mean compressibility value over 5 consecutive measurements. Malignancy ground truth will be defined based on standard of care post-surgical histopathological results.

CONTACTS AND LOCATIONS:
Overall Officials: PD Dr. med. Urs Borner, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Department of Oto-Rhino-Laryngology, Head and Neck surgery Inselspital, Bern University Hospital and University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No